## The GlaxoSmithKline group of companies

204745

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for 204745: An open-label, single arm study to investigate the safety, pharmacokinetics and pharmacodynamics of repeat doses of inhaled GSK2269557 in patients with APDS/PASLI |
| <b>Compound Number</b> | : | GSK2269557 |
| <b>Effective Date</b> | : | Refer to Document Date |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 204745.
- This RAP is intended to describe the final analyses required for the study.
- This version of the RAP includes amendments to the originally approved Critical Components of the RAP.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

# **RAP Author(s):**

| Author | |
|---|---|
| PPD | |
| Principal Statistician (Clinical Statistics) | |
| PPD | |
| Associate Sta | atistician (Clinical Statistics) |

Copyright 2021 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

The GlaxoSmithKline group of companies

204745

## **RAP Team Reviews:**

# **RAP Team Review Confirmations**

(Method: E-mail)

| Reviewer | Date |
|---|---|
| Global Clinical Development Manager (Respiratory Global Clinical Sciences and Discovery) | 15-DEC-2020 |
| Early Discovery Lead<br>(Respiratory Early Discovery Leaders) | 19-NOV-2020 |
| Sr Director Clinical Pharmacology (Respiratory Clinical Pharmacology Modelling and Simulation) | 28-NOV-2020 |
| Discovery Medicine Physician Director (Discovery Medicine) | 17-DEC-2020 |
| Programming Leader (Respiratory, Clinical Programming) | 26-NOV-2020 |

# **Clinical Statistics and Clinical Programming Line Approvals:**

# **Clinical Statistics & Clinical Programming Line Approvals**

(Method: Veeva Clinical Vault eSignature)

| Approver |
|-------------------------------------|
| PPD |
| Statistics Director |
| (Respiratory, Clinical Statistics) |
| PPD |
| Programming Director |
| (Respiratory, Clinical Programming) |

204745

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | DUCTION | | 6 |
| 2. | SLIMM | ABA UE KE | EY PROTOCOL INFORMATION | 6 |
| ۷. | | | the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Obje | ective(s) and Endpoint(s) | 7 |
| | | | gn | |
| | | | Hypotheses / Statistical Analyses | |
| 3. | | | 'SES | |
| | | | alyses | |
| | 3.2. | Final Analy | ses | 10 |
| 4. | ANALY | SIS POPU | LATIONS | 10 |
| | 4.1. | Protocol De | eviations | 10 |
| _ | CONOL | DEDATION | IO FOR DATA ANALYOFO AND DATA HANDLING | |
| 5. | | | IS FOR DATA ANALYSES AND DATA HANDLING | 12 |
| | | | tment & Sub-group Display Descriptors | |
| | | | efinitions | |
| | - | | siderations for Data Analyses and Data Handling | |
| | | Convention | 18 | 14 |
| | O.T. I.D. | | | |
| 6. | | | TION ANALYSES | |
| | 6.1. | Overview o | of Planned Study Population Analyses | 15 |
| 7. | SAFET | Y ANALYS | ES | 16 |
| | 7.1. | Adverse Ev | vents Analyses | 16 |
| | 7.2. | Clinical Lab | poratory Analyses | 16 |
| | 7.3. | Other Safe | ty Analyses | 16 |
| 8. | PHARI | 1ACOKINE | TIC ANALYSES | 17 |
| ٥. | | | Pharmacokinetic Analyses | |
| | | | Indpoint / Variables | |
| | | | .1.1.1. Drug Concentration Measures | |
| | | | .1.1.2. Derived Pharmacokinetic Parameters | |
| | | 8.1.2. S | ummary Measure | |
| | | | opulation of Interest | |
| | | | trategy for Intercurrent Events | |
| | | 8.1.5. S | statistical Analyses / Methods | 17 |
| | 8.2. | Exploratory | / Pharmacokinetic Analyses | 18 |
| | | | indpoint / Variables | |
| | | 8 | .2.1.1. Drug Concentration Measures | 18 |
| | | | .2.1.2. Derived Pharmacokinetic Parameters | |
| | | | summary Measure | |
| | | | opulation of Interest | |
| | | 8.2.4. S | trategy for Intercurrent Events | 18 |
| | | 8.2.5. S | tatistical Analyses / Methods | 19 |
| ۵ | | ΙΔΟΟΠΥΝΙ | AMIC AND BIOMARKER ANALYSES | 20 |

204745

9.1. 9.1.1. 9.1.2. Summary Measure ......20 9.1.3. 9.1.4. 9.1.5. Statistical Methodology Specification......21 10.1.1. 10.1.3. 10 1 4 11. REFERENCES 23 Appendix 1: Protocol Deviation Management .......24 12.2. Appendix 3: Study Phases and Treatment Emergent Adverse 12.3. 12.3.1. 12.3.1.1. Study Phases for Concomitant Medication .......30 12.3.2. 12.3.3. 12.4. 12.4.1. Reporting Standards 32 12.4.2. 12.4.3. 12.5. 12.5.1. General 34 12.5.2. 12.5.3. 12.5.4. 12.5.5. 12.5.6. 12.6. Appendix 6: Reporting Standards for Missing Data......39 12.6.1. 12.6.2. Handling of Missing Data ......39 12.6.2.1. Handling of Missing and Partial Dates ...............................40 12.7. Laboratory Values.......42 12.7.1. 12.7.2. Vital Signs......43 12.7.3. 12.8. Appendix 9: Abbreviations & Trade Marks .......45 12.9. Abbreviations .......45 12.9.2. 12.10. Appendix 10: List of Data Displays......47 

| | 204745 |
|-----------------------------------------------------------|--------|
| 12.10.3. Deliverables | 47 |
| 12.10.4. Study Population Tables | 48 |
| 12.10.5. Efficacy Tables | 49 |
| 12.10.6. Safety Tables | 50 |
| 12.10.7. Pharmacokinetics Table | |
| 12.10.8. Pharmacodynamic and Biomarker Tables | 52 |
| 12.10.9. Pharmacodynamic and Biomarker Figures | 53 |
| 12.10.10.ICH Listings | 54 |
| 12.10.11.Non-ICH Listings | |
| 12.11. Appendix 11: Example Mock shells for Data Displays | |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| 2015N238311_00 | 23-OCT-<br>2015 | Original |
| 2015N238311_01 | 25-FEB-2016 | Amendment No. 1 [Update to include modification requested by MHRA to extend the duration of contraception after end of study} |
| 2015N238311_02 | 02-<br>NOV_2016 | Amendment No. 2 [To change IMP device from Diskus to Ellipta] |
| 2015N238311_03 | 15-JUN-2017 | Amendment No. 3 [New formulation GSK2269557 will be administered via the ELLIPTA™ dry powder inhaler (DPI) formulated in a blend containing 0.4% MgSt (magnesium stearate). The previous formulation contained 0.6% MgSt.] |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| The exploratory endpoints specified in Protocol amendment 3 were: Endpoints may include, but are not limited to: In blood and sputum, analysis of: • Cellular PIP3 peak area as a proportion of (PIP3 peak area + PIP2 peak area) • Soluble proinflammatory mediators (including IL-8, IL-6, TNFα & MMP9) • Immune cell subsets • Exploratory phospho-protein biomarkers (e.g. pAKT) • Exploratory messenger ribonucleic | The exploratory endpoints specified in this RAP are: Endpoints may include, but are not limited to: In blood and sputum, analysis of: • Cellular PIP3 peak area as a proportion of (PIP3 peak area + PIP2 peak area) • Soluble proinflammatory mediators (including IL-8, IL-6, TNFα & MMP9) • Immune cell subsets (In Sputum only) • Lymphocyte cell subsets • Exploratory phospho-protein biomarkers (e.g. pAKT) | Exploratory mRNA biomarkers (in blood, sputum, BAL cell pellet/lavage supernatant); proteomic markers (in lavage supernatant) and bacterial DNA fragments (in blood) analysis were not conducted. As a result, they have been removed from the RAP. |
| acid (mRNA) biomarkers In BAL cell pellet/lavage supernatant when available, analysis of: Lymphocyte cell subsets | <ul> <li>Antibody levels</li> <li>In BAL cell pellet/lavage supernatant when available, analysis of:</li> <li>Lymphocyte cell subsets</li> </ul> | |

204745

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| <ul> <li>Exploratory phospho-protein biomarkers (e.g. pAKT)</li> <li>Soluble proinflammatory mediators (including IL-8, IL-6, TNFα &amp; MMP9)</li> <li>Exploratory mRNA biomarkers</li> <li>Proteomic markers (lavage supernatant only)</li> <li>Antibody levels</li> <li>In blood, analysis of:</li> <li>Bacterial DNA fragments</li> </ul> | <ul> <li>Exploratory phospho-protein biomarkers (e.g. pAKT)</li> <li>Immune cell subsets</li> <li>Soluble proinflammatory mediators (IL-8, IL-6, TNFα &amp; MMP9)</li> </ul> | |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| Safety • To assess the safety and tolerability of 84 days repeat dosing of inhaled nemiralisib in patients with APDS | <ul> <li>Adverse Events (AE)</li> <li>Vital signs</li> <li>12-lead electrocardiogram (ECG)</li> <li>Clinical laboratory parameters</li> <li>Spirometry (forced expiratory volume in 1 second (FEV1)1 hr post-dose)</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| <ul> <li>Pharmacokinetics</li> <li>To define the plasma pharmacokinetics (PK) of inhaled nemiralisib following repeat dosing in patients with APDS.</li> </ul> | <ul> <li>Nemiralisib trough plasma concentration following<br/>single and repeated treatment.</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| Pharmacodynamics: To understand lung disease biology in patients with APDS and to explore the pharmacodynamic effects of inhaled nemiralisib. | <ul> <li>Endpoints may include, but are not limited to:</li> <li>In blood and sputum, analysis of:</li> <li>Cellular PIP3 peak area as a proportion of (PIP3 peak area + PIP2 peak area)</li> <li>Soluble proinflammatory mediators (IL-8, IL-6, TNFα &amp; MMP9)</li> <li>Immune cell subsets (In Sputum Only)</li> <li>Lymphocyte cell subsets</li> <li>Exploratory phospho-protein biomarkers (e.g. pAKT)</li> <li>Antibody Levels</li> </ul> |
| | In BAL cell pellet/lavage supernatant when available, analysis of: |
| | <ul> <li>Lymphocyte cell subsets</li> <li>Exploratory phospho-protein biomarkers (e.g. pAKT)</li> <li>Immune cell subsets</li> </ul> |

204745

| Objectives | Endpoints |
|---|---|
| | • Soluble proinflammatory mediators (including IL-8, IL-6, TNFα & MMP9) |
| Pharmacokinetics: To define the lung trough concentration of nemiralisib after repeat dosing | Trough nemiralisib concentration in lung epithelial lining fluid (ELF) and Bronchoalveolar lavage (BAL) cell pellet at Day 84 visit. |
| <ul> <li>Efficacy:</li> <li>To assess the efficacy of inhaled</li> <li>nemiralisib administered once daily for 84 days in patients with APDS.</li> </ul> | <ul> <li>The number and rate of pulmonary and/or ear and sinus infections requiring anti-microbial treatment compared to subject's historical baseline.</li> <li>Change from baseline (Day 1) in trough FEV1 at Day 14 and Day 83 (prebronchodilator)</li> </ul> |

# 2.3. Study Design



# 2.4. Statistical Hypotheses / Statistical Analyses

No formal statistical hypotheses will be tested.

## 3. PLANNED ANALYSES

# 3.1. Interim Analyses

Formal interim analyses will not be performed. However, safety, pharmacokinetic and pharmacodynamic data will be reviewed on an ongoing basis for internal decision-making purposes, to ensure subject safety and to maximise the ability to measure multiple PD markers based on sample availability.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | <ul> <li>All participants who were screened for eligibility</li> <li>This population will be based on the treatment the subject received.</li> <li>If participants receive no treatment, then they will be summarised according to "No Treatment"</li> </ul> | Study Population |
| All Subjects | <ul> <li>All subjects who receive at least one dose of the study treatment.</li> <li>This population will be based on the treatment the subject received.</li> </ul> | <ul><li>Study Population</li><li>Safety</li><li>Efficacy</li><li>PD/Biomarker</li></ul> |
| Pharmacokinetic<br>(PK) | <ul> <li>All participants in the 'All Subjects' population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values).</li> <li>This population will be based on the treatment the subject received.</li> <li>Note: PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded.</li> </ul> | • PK |

Refer to Appendix 10: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

204745

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan Version2.0 [19/Feb/2019].

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A listing of all inclusion/exclusion criteria deviations will be provided. This will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description | Order in TLF |
| Α | GSK2269557 1000 mcg | NEMI 1000mcg Diskus | 1 |
| В | GSK2269557 700 mcg | NEMI 700mcg Ellipta | 2 |
| С | Nemiralisib 500 mcg | NEMI 500mcg Ellipta | 3 |
| This will be codes A/B | e derived as subjects in RandALL<br>//C | All NEMI | 4 |
| | e derived as subjects who did not<br>ny treatment | No Treatment | 5 |

#### Note:

- Due to the protocol amendments subjects may have been assigned to Nemiralisib 1000 μg via the Diskus device, Nemiralisib 700 μg via the Ellipta device or Nemiralisib 500 μg via the Ellipta device depending on the protocol amendment they were enrolled on. These treatments were intended to be comparable hence the "All NEMI" Treatment group will be created.
- Pharmacodynamic and Biomarker, Efficacy and study population (except exposure summary) domain summaries will be presented for "All NEMI" Treatment group only.
- "NEMI 1000mcg Diskus" / "NEMI 700mcg Ellipta" / "NEMI 500mcg Ellipta" treatment groups will be presented in PK domain and all listings.
- "NEMI 1000mcg Diskus" / "NEMI 700mcg Ellipta"/ "NEMI 500mcg Ellipta" and "All NEMI" treatment groups will be presented in Safety Domain summaries and Exposure Summary Tables.

204745

## 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study A | ssessmei<br>Bas | lered as | Baseline Used in<br>Data Display | |
|---|---|---|---|---|---|
| | Screening | Clinic<br>Visit 1 | Day -1 | Day 1<br>(Pre-<br>Dose) | |
| Efficacy | | | | | • |
| FEV1 <sup>1</sup> | Х | | | Х | Day 1 (Pre dose) |
| Ear, sinus and pulmonary infection history | Х | | | | Screening |
| Safety | | | | | • |
| Vital signs | Χ | Х | Х | Χ | Day 1 (Pre dose) |
| 12-lead ECG | Χ | Χ | Χ | Χ | Day 1 (Pre dose) |
| Spirometry | Χ | | | Χ | Day 1(Pre dose) |
| Laboratory assessments | Χ | Х | Х | | Day -1 |
| Pharmacodynamic and Biomarker | S | | | | |
| PD blood sample <sup>2</sup> | | Χ | Χ | | Day -1 |
| BAL sub-study only:<br>Bronchoscopy/BAL | | Х | | | Clinic Visit 1<br>(At least 7 days<br>prior to dosing) |
| BAL sub-study only: Additional haematology Assessments <sup>3</sup> | | Х | | _ | Clinic Visit 1<br>(At least 7 days<br>prior to dosing) |

<sup>1 –</sup> prebronchodilator

<sup>2 -</sup> PD blood sample to include, but not limited to Lymphocyte assessments, PIP2/PIP3 assessments, soluble proinflammatory mediators

<sup>3 -</sup> For clotting status (Activated partial thromboplastin time (aPTT), Prothrombin time (PT))

204745

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 12.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 12.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 12.5 | Appendix 5: Derived and Transformed Data |
| 12.6 | Appendix 6: Reporting Standards for Missing Data |
| 12.7 | Appendix 7: Values of Potential Clinical Importance |

204745

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "All Subjects" population, unless otherwise specified.

Study population analyses, including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance, will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

204745

## 7. SAFETY ANALYSES

The safety analyses will be based on the "All Subjects" population, unless otherwise specified.

# 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

## 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 10: List of Data Displays.

## 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 10: List of Data Displays.

## 8. PHARMACOKINETIC ANALYSES

## 8.1. Secondary Pharmacokinetic Analyses

## 8.1.1. Endpoint / Variables

• Nemiralisib plasma concentration

## 8.1.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 12.4.3 Reporting Standards for Pharmacokinetic)

#### 8.1.1.2. Derived Pharmacokinetic Parameters

No pharmacokinetic parameters will be calculated. concentration measured 24 hours post-dose/pre-dose are assumed to be trough concentrations.

## 8.1.2. Summary Measure

The geometric mean of Nemiralisib plasma concentration following single (Day 1: Predose, 5 min, 3 h and 24 h post-dose) and repeated treatment (Day 14 Pre-dose, Day 83 Pre-dose and Early withdrawal) will be summarised for the treatment groups: "NEMI 1000mcg Diskus", "NEMI 700mcg Ellipta" and "NEMI 500mcg Ellipta". Flag will be derived to see whether values range fall within the 2-fold range to check data decision framework as detailed in Section 12.8

## 8.1.3. Population of Interest

The plasma pharmacokinetic summaries will be based on the "Pharmacokinetic" population.

## 8.1.4. Strategy for Intercurrent Events

Intercurrent events have been considered e.g. discontinuation of treatment and treatment switching. Due to the exploratory nature of this study and small sample size we accept these intercurrent events may have an impact on the endpoints which we are unable to quantify. Therefore, a treatment policy approach will be adopted hence the actual values of the endpoint, regardless of whether the intercurrent event has occurred, will be analysed.

# 8.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics and listed.

## 8.2. Exploratory Pharmacokinetic Analyses

## 8.2.1. Endpoint / Variables

Nemiralisib concentration in lung epithelial lining fluid (ELF) and Bronchoalveolar lavage (BAL) cell pellet at Day 84 visit.

## 8.2.1.1. Drug Concentration Measures

Lung epithelial lining fluid (ELF) and BAL cell pellet analysis for nemiralisib will be performed under the management of PTS-DMPK, GlaxoSmithKline. Concentrations of nemiralisib will be determined using the currently approved bioanalytical methodology.

## 8.2.1.2. Derived Pharmacokinetic Parameters

No lung pharmacokinetic parameters will be calculated; concentration measured 24 hours post-dose/pre-dose are assumed to be trough concentrations.

## 8.2.2. Summary Measure

The geometric mean of Nemiralisib concentration in the lung epithelial lining fluid (ELF) and Bronchoalveolar lavage (BAL) cell pellet at Day 84 visit will be summarised for the treatment groups: "NEMI 1000mcg Diskus", "NEMI 700mcg Ellipta" and "NEMI 500mcg Ellipta".

- BAL fluid and plasma urea data, along with the derived Dilution Factor (see Section 12.5.4 for derivation) for each wash, will be listed. See Section 12.6.2 for the handling of BLQ values when calculating the Dilution Factor
- BAL fluid concentrations of GSK2269557 and derived ELF concentrations of GSK2269557 (corrected for by Dilution Factor) for each wash will be listed. In addition, volumes of ELF and the amount of GSK2269557 in the BAL fluid sample will be included in the listing, in order to derive the pooled ELF concentration of GSK2269557 (across all the washes). All applicable derivations are detailed in Section 12.5.4

## 8.2.3. Population of Interest

The lung pharmacokinetic summaries will be based on the "Pharmacokinetic" population.

## 8.2.4. Strategy for Intercurrent Events

Intercurrent events have been considered e.g. discontinuation of treatment, treatment switching and death. Due to the exploratory nature of this study and small sample size we accept these intercurrent events may have an impact on the endpoints which we are unable to quantify. Therefore, a treatment policy approach will be adopted hence the actual values of the endpoint regardless of whether the intercurrent event has occurred will be analysed.

204745

# 8.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics and listed.

## 9. PHARMACODYNAMIC AND BIOMARKER ANALYSES

## 9.1. Exploratory Pharmacodynamic and Biomarker Analyses

## 9.1.1. Endpoint / Variables

Endpoints may include, but are not limited to:

#### In blood and sputum, analysis of:

- Cellular PIP3 peak area as a proportion of (PIP3 peak area + PIP2 peak area)
- Soluble proinflammatory mediators (IL-8, IL-6, TNFα & MMP9)
- Immune cell subsets (In Sputum Only)
- Lymphocyte cell subsets
- Exploratory phospho-protein biomarkers (e.g. pAKT)
- Antibody Levels

## In BAL cell pellet/lavage supernatant when available, analysis of:

- Lymphocyte cell subsets
- Exploratory phospho-protein biomarkers (e.g. pAKT)
- Immune cell subsets
- Soluble proinflammatory mediators (including IL-8, IL-6, TNFα & MMP9)

## 9.1.2. Summary Measure

Absolute and Change from Baseline/Ratio to Baseline will summarised using descriptive statistics for each timepoint as defined in Section 9.1.1

## 9.1.3. Population of Interest

The pharmacodynamics analyses will be based on the "All Subjects" population, unless otherwise specified.

## 9.1.4. Strategy for Intercurrent Events

Several intercurrent events have been considered e.g. infections, use of rescue medication, discontinuation of treatment, treatment switching and death. Due to the exploratory nature of this study and small sample size we accept these intercurrent events may have an impact on the endpoints which we are unable to quantify. Therefore, a treatment policy approach will be adopted hence the actual values of the endpoint regardless of whether the intercurrent event has occurred will be analysed.

## 9.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

204745

## 9.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Loge-transformed PIP3 Area Proportion

## **Model Specification**

- will be analyzed using mixed models repeated measures (MMRM) models for Blood Sample Type.
- Terms fitted in the model will include:
  - Fixed Effect: Processing Type, Visit
  - Random Effect: Subject
  - Repeated: Visit

Note: Per the analysis population all subjects will be within the "All NEMI" treatment group and as such treatment arm need not be included as a fixed effect in the model

- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
- In the event that this model fails to converge, the estimates will not be reported.
- Point estimates for the adjusted means on the loge scale, the mean ratio between processing
  Type and associated 95% confidence interval will be constructed using the residual variance
  for the following combination of interest:
  - Unstimulated+DMSO / Stimulated+DMSO
  - Unstimulated+DMSO / Unstimulated+NEMI
  - Stimulated+DMSO / Stimulated+NEMI

## **Model Checking & Diagnostics**

Distributional assumptions underlying the model used for analysis will be examined by
obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
values (i.e. checking the normality assumption and constant variance assumption of the
model respectively) to gain confidence that the model assumptions are reasonable.

#### **Model Results Presentation**

- The point estimate and confidence interval obtained from MMRM analysis will be exponentially back-transformed to obtain Adjusted (least square) geometric means for each processing type
- The adjusted mean ratio and associated 95% confidence interval for the following processing type combinations:
  - Unstimulated+DMSO / Stimulated+DMSO
  - Unstimulated+DMSO / Unstimulated+NEMI
  - Stimulated+DMSO / Stimulated+NEMI

## 10. EFFICACY ANALYSES

# 10.1. Exploratory Efficacy Analyses

## 10.1.1. Endpoint / Variables

- Pulmonary and/or ear and sinus infections requiring anti-microbial treatment, refer to Section 12.5.6. for how these will be programmatically identified.
- FEV1

## 10.1.2. Summary Measure

The number and rate (per 84 days) of pulmonary and/or ear and sinus infections requiring anti- microbial treatment will be calculated for each subject.

Mean change from baseline FEV1 at Day 14:pre-dose, Day 83:pre-dose, early withdrawal and 3 month follow up will be summarised for the "All NEMI" treatment group.

## 10.1.3. Strategy for Intercurrent Events

Several intercurrent events have been considered e.g. infections, use of rescue medication, discontinuation of treatment, treatment switching and death. Due to the exploratory nature of this study and small sample size we accept these intercurrent events may have an impact on the endpoints which we are unable to quantify. Therefore, a treatment policy approach will be adopted hence the actual values of the endpoint regardless of whether the intercurrent event has occurred will be analysed.

## 10.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.1.1 will be listed.

204745

# 11. REFERENCES

GlaxoSmithKline Document Number 2012N141231\_10. Nemiralisib (GSK2269557) Investigator's Brochure: 03-AUG-2018

GlaxoSmithKline Document Number 2015N238311\_03. An open-label, single arm study to investigate the safety, pharmacokinetics and pharmacodynamics of repeat doses of inhaled nemiralisib in patients with APDS/PASLI 30-MAY-2017

204745

# 12. APPENDICES

# 12.1. Appendix 1: Protocol Deviation Management

Instream and final analysis population reviews as per SOP 130050 will be conducted. Please Refer to Section 4.1 for handling and Reporting of Protocol Deviations.

204745

# 12.2. Appendix 2: Schedule of Activities

# Time and Events Table for Screening and Run-in Period

| Procedure | Pre-<br>Screening | Screening | Clinic visit #1 | Notes |
|---|---|---|---|---|
| | | (up to 42 days prior to dosing) | At least 7 days prior to dosing | |
| Informed consent | X | | | Pre-screening and screening may occur on the same visit,<br>if appropriate |
| Concomitant medication review | X | | | |
| Review of exacerbation<br>history | X | | | |
| Demography | X | X | | |
| SAE review | X | X | X | |
| Inclusion and exclusion<br>criteria | | X | | |
| Full physical exam, including<br>height and weight | | X | | |
| Brief physical examination | | | X | |
| Medical history (includes<br>substance usage and Family<br>history of premature CV<br>disease) | | X | | Substances: Drugs, Alcohol, tobacco |
| Past and current medical<br>conditions (including ear,<br>sinus and pulmonary<br>infection history,<br>cardiovascular medical<br>history and therapy history) | | X | | |
| Vital signs (Blood pressure<br>(BP), heart rate (HR),<br>temperature and respiratory<br>rate) | | Х | Х | Triplicate measurements of BP and HR |
| 12-lead ECG | | X | X | Triplicate |

204745

| Procedure | Pre-<br>Screening | Screening | Clinic visit #1 | Notes |
|---|---|---|---|---|
| | 17 | (up to 42 days prior to dosing) | At least 7 days prior to dosing | |
| Spirometry (incl. reversibility) | | X | | |
| Laboratory assessments<br>(include hematology,<br>biochemistry, Urinalysis) | | Х | Х | |
| HIV, Hep B and Hep C<br>screen | | X | | |
| Blood pregnancy test (only WCBP) | | Х | | |
| PD blood sample:<br>Lymphocyte assessments<br>(subset counts, soluble<br>proinflammatory mediators,<br>phosphoprotein biomarkers,<br>immunoglobulins.) | | | X | |
| PD blood sample: PIP <sub>2</sub> /PIP <sub>3</sub><br>assessments | | | Х | |
| PD blood sample: mRNA<br>biomarkers | | | Х | |
| PD blood sample: bacterial<br>DNA fragment analysis | | | Х | |
| Sputum induction | | | Х | Should sputum induction fail or be insufficient, the subject will be allowed to return within 48 hours for a further attempt to obtain an adequate sample |
| BAL sub-study only:<br>Bronchoscopy/BAL | | | Х | Performed on a different day to the sputum induction.<br>For measurement of PD |
| BAL sub-study only:<br>Additional haematology<br>assessments | | | Х | For clotting status (Activated partial thromboplastin time (aPTT), Prothrombin time (PT)) |

204745

# Time and Events Table for Treatment Period and Follow-up

| Procedure | | Treatment Period | | | | | | | | | | w-up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Clinic Visit | | 2 | | 3 | | 4 | 5 | ( | ô | Early | 1-2 | 7 | |
| Day | -1 | 1 | 2 | 14 | 2 to<br>84 | 28 | 56 | 83 | 84‡ | with-<br>drawal | wks | 3 mths | Notes |
| Visit window | N/A | N/A | N/A | ±2<br>days | ±3<br>days | -4 / +2<br>days | -4 / +2<br>days | -4 / +2<br>days | -4 / +2<br>days | (within<br>2 wks) | 4-6 | ±2<br>weeks | |
| In-Patient | Х | X | Х | | | | | | | | | | |
| Out-Patient | | | | Х | | Х | Х | Х | Х | Х | | Х | |
| Telephone Contact/<br>Research nurse visit | | | | | X<br>weekly | | | | | | Х | | Except weeks where subjects have a clinic visit |
| | | | | | | SAFE | TY AS | SESSM | ENTS | | | | |
| Brief physical exam | Х | | | Х | | Х | Х | Х | | Х | | Х | Pre-dose |
| AE/SAE review | ←== | | | | | | | | | <i>&gt;</i> | Х | Х | |
| Concomitant medication review | ←== | | | | | | | | | ===→ | Х | Х | |
| Vital signs | Х | Х | | Х | | Х | Х | Х | Х | Х | | Х | Pre-dose. Single assessment |
| 12-lead ECG | Х | Х | | Х | | Х | Х | Х | | Х | | Х | Pre-dose. Single assessment |
| Urine pregnancy test | Х | | | Х | | | Х | Х | | Х | | | only WCBP |
| Laboratory assessments (include<br>haematology, biochemistry,<br>Urinalysis) | х | | | х | | х | х | х | | Х | | х | Pre-dose |
| | | | | | | ST | UDY TR | EATME | NT | | | | |
| ELLIPTA inhaler training | х | | | | | | | | | | | | Review of the Patient Information Leaflet with the<br>subject (no device will be used). Additional training<br>may be conducted at the discretion of the<br>investigator |
| Study drug administration | | < | | | | | | | | | | | Daily in the morning before breakfast, (with the<br>exception of days when the subjects have a<br>planned visit to the clinic. On those days, they will |

| Procedure | | | | Т | reatme | nt Perio | od | | | | | w-up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Clinic Visit | | 2 | | 3 | | 4 | 5 | 6 | i | Early | 1-2 | 7 | |
| Day | -1 | 1 | 2 | 14 | 2 to<br>84 | 28 | 56 | 83 | 84‡ | with-<br>drawal | wks<br>and | 3 mths | Notes |
| Visit window | N/A | N/A | N/A | ±2<br>days | ±3<br>days | -4 / +2<br>days | -4 / +2<br>days | -4 / +2<br>days | | (within<br>2 wks) | 4-6<br>wks | ±2<br>weeks | |
| In-Patient | Х | Х | Χ | | | | | | | | | | |
| Out-Patient | | | | X | | Х | Х | Х | X | Х | | Х | |
| Telephone Contact/<br>Research nurse visit | | | | | X<br>weekly | | | | | | Х | | Except weeks where subjects have a clinic visit |
| | | | | | | | | | | | | | be dosed at the clinic). |
| Assessment of study treatment compliance | | | | X | | Х | Х | Х | | х | | | |
| | | | | | | EFFIC. | ACY AS | SESSN | IENTS | | | | |
| Exit interview | | | | | | | | Х | | x | | | Exit interview may be held at the study clinic or the<br>subject's home, within 7 days of last dose. |
| | | | | | | OTH | ER ASS | ESSME | NTS | | | | |
| Review of APDS exacerbation and<br>respiratory tract infection history | | | | X | | X | х | Х | | X | Х | Х | Including ear, sinus and pulmonary infections. |
| FEV1 Pre-Dose | | Х | | X | | | | Х | | X | | Х | For efficacy |
| FEV1 1hr Post-Dose | | Х | Х | Х | | | | | | | | | For safety |
| Blood sample for PK | | Х | | Х | | | | х | | Х | | | Day 1: Pre-dose, 5 min, 3 h and 24 h post-dose.<br>Pre-dose at all other visits. |
| PD blood sample: Lymphocyte assessments | x | | | X | | | | х | | х | | | Pre-dose. Subset counts, soluble proinflammatory<br>mediators, phosphoprotein biomarkers,<br>immunoglobulins. |
| PD blood sample: PIP <sub>2</sub> /PIP <sub>3</sub> assessments | х | | | Х | | | | х | | Х | | Х | Pre-dose. |

204745

| Procedure | | Treatment Period | | | | | | | | | Follow-up<br>Period | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Clinic Visit | | 2 | | 3 | | 4 | 5 | ( | 3 | Early | 1-2 | 7 | |
| Day | -1 | 1 | 2 | 14 | 2 to<br>84 | 28 | 56 | 83 | 84‡ | with-<br>drawal | wks<br>and | 3 mths | Notes |
| Visit window | N/A | N/A | N/A | ±2<br>days | ±3<br>days | -4 / +2<br>days | -4 / +2<br>days | -4 / +2<br>days | -4 / +2<br>days | (within<br>2 wks) | 4-6<br>wks | ±2<br>weeks | |
| In-Patient | Х | Х | X | | | | | | | | | | |
| Out-Patient | | | | Х | | Х | Х | Х | Х | X | | X | |
| Telephone Contact/<br>Research nurse visit | | | | | X<br>weekly | | | | | | Х | | Except weeks where subjects have a clinic visit |
| PD blood sample: mRNA biomarkers | Х | | | х | | | | X | | х | | х | Pre-dose. |
| PD blood sample: bacterial DNA<br>fragment analysis | Х | | | Х | | | | X | | Х | | | Pre-dose. |
| Sputum induction | х | | | х | | | | х | | | | х | Pre-dose. Should sputum induction fail or be<br>insufficient, the subject will be allowed to return<br>within 48 hours for a further attempt to obtain an<br>adequate sample |
| BAL sub-study only: Additional<br>haematology assessments | | | | | | | | X | | | | | For clotting status (Activated partial thromboplastin<br>time (aPTT), Prothrombin time (PT)) |
| BAL sub-study only:<br>Bronchoscopy/BAL | | | | | | | | | x | | | | For measurement of PK and PD |
| BAL sub-study only:<br>Blood sample for urea PK | | | | | | | | | х | | | | |
| BAL sub-study only:<br>Blood sample for plasma PK | | | | | | | | | х | | | | |
| Genetic Sample | х | | | | | | | | | | | | Optional assessment – the subject must provide<br>additional consent for the genetic sample. Genetic<br>sample can be taken at any time after<br>randomisation. |

<sup>‡</sup> Day 84 visit will only occur if a subject has agreed to take part in the BAL sub-study, dosing will continue until the D84 visit.

204745

# 12.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

# 12.3.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment start date.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date |
| Post-Treatment | atment Date > Study Treatment Stop Date |
| NOTES: | |
| Time of study treat collected. | atment dosing and start/stop time of assessments and events should be considered, if |

## 12.3.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

• Please refer to Appendix 6: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

#### 12.3.2. Treatment States for Adverse Events

| Flag | Definition |
|---|---|
| Pre-Treatment | If AE onset date is before the treatment start date. |
| | AE Start Date < Study Treatment Start Date |
| Treatment<br>Emergent | If AE onset date is on or after treatment start date & on or before treatment stop date. |
| (On-Treatment) | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date. |
| Post-Treatment | If AE onset date is after the treatment stop date. |
| | AE Start Date > Study Treatment Stop Date |

## NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

204745

# 12.3.3. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date is on or after treatment start date &amp; on or before treatment stop date.</li> <li>Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date</li> </ul> |

## NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

204745

# 12.4. Appendix 4: Data Display Standards & Handling Conventions

# 12.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software (version 9.4) will be used. | |
| Reporting Area | |
| HARP Server | : UK1SALX00175.corpnet2.com |
| HARP Compound | : ARPROD/GSK2269557/mid204745 |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK A&R dataset standards and Integrated Data Standards Library | |
| Generation of RTF Files | |
| RTF files will be generated for all tables | |

## 12.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings
- A project wide decision was made to present GSK2269557 as Nemiralisib (abbreviated to NEMI) refer to Section 5.1 for further details.

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

## **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

204745

| Unscheduled Visits | |
|---|---|
| Unscheduled visits will not be included in summary tables and/or figures | |
| All unscheduled visits will be included in listings. | |
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 12.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| Descriptive | Refer to IDSL PK Display Standards. |
| Summary Statistics, | Refer to IDSL Statistical Principle 6.06.1. |
| Graphical Displays | Note: Concentration values will be imputed as per GUI_51487 for descriptive |
| and Listings | summary statistics/analysis and summarized graphical displays only. |
| | Note: Use the separate NEMI DISKUS and NEMI ELLIPTA treatment groups |

204745

## 12.5. Appendix 5: Derived and Transformed Data

#### 12.5.1. General

#### Multiple Measurements at One Analysis Time Point

Where multiple measurements are recorded for a particular time point, all available data will be listed. The mean of the measurements will be calculated and used in the derivation of summary statistics; except in the following cases:

- FEV1 data: in the calculation of summary statistics, the maximum of triplicate readings will be used
- Biomarker data: in the calculation of summary statistics/for statistical analyses, assuming the data appears log normally distributed, the geometric mean of the two replicates will be used.

If there are two values within a protocol scheduled visit the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.

Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

## Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

# 12.5.2. Study Population

## **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age at Screening where birth date will be imputed as follows:
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Refer to IDSL standards for age range categories.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)^2]

#### **Extent of Exposure**

• Number of days of exposure to study drug will be calculated based on the formula:

### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Participants who were assigned a treatment but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### **Cumulative Dose = Sum of (Counter Readings x Container Dose)**

If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

204745

## 12.5.3. Safety

## **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Decimal Places = '< x ' becomes x 0.01
  - Example 2: 1 Decimal Place = '> x' becomes x + 0.1
  - Example 3: 0 Decimal Places = '< x' becomes x 1

#### **ECG Parameters**

#### **RR Interval**

IF RR interval (msec) is not provided directly, then RR can be derived as:
 [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value then
do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as:

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### 12.5.4. Pharmacokinetic

#### **ELF Drug Concentrations**

Urea concentration data in plasma and BAL will be used to calculate the dilution effect of the lavage which is used to extract the epithelial lining fluid (ELF) from the lung compartment. A correction for dilution will be applied to all BAL analytes to derive corrected concentrations i.e. each BAL analyte will be adjusted to account for the magnitude of dilution during the BAL procedure using urea plasma concentration as a reference point. A correction for dilution will be applied to all BAL fluid drug concentrations for each wash as follows:

ELF Concentration 
$$(pg/ml)$$
  
= BAL Drug Concentration  $(pg/ml) * Dilution Factor$ 

Where

204745

$$Dilution Factor = \frac{Urea \ Plasma \ _{pre-bronch}}{Urea \ BAL}$$

Additionally, for each wash, the Volume of ELF in BAL fluid and the Total Drug in BAL fluid will be calculated as follows:

Volume of ELF in BAL Fluid (mL) = 
$$\frac{BAL \ Fluid \ Volume \ (mL)}{Dilution \ Factor}$$

Drug in BAL Fluid (pg) = BAL Fluid Drug Concentration  $(\frac{pg}{mL}) * BAL$  Fluid Volume (mL)

Data will then be pooled across all three washes as follows:

 $Total\ Drug\ in\ BAL\ Fluid\ (pg) = Drug\ in\ BAL_{wash1} + Drug\ in\ BAL_{wash2} + Drug\ in\ BAL_{wash3}$ 

Pooled ELF Drug Concentration 
$$\left(\frac{pg}{mL}\right) = \frac{Total\ Drug\ in\ BAL\ Fluid\ (pg)}{Total\ Volume\ of\ ELF\ in\ BAL\ Fluid\ (mL)}$$

## **BAL Cell Pellet Drug Concentration**

Cell pellet samples are diluted in a 1:5 ratio. Concentrations will be corrected for the dilution before the ratio is calculated on an individual subject level between the raw lavage result for wash 2 and the cell pellet concentration:

 $\label{eq:definition} \begin{aligned} & \textit{Derived cell pellet concentration} \\ & = \frac{\textit{cell pellet concentration} * 5}{\textit{wash 2 lavage concentration}} * \textit{derived pooled lavage ELF concentration} \end{aligned}$ 

Only the derived concentrations will be included in the listing.
204745

#### 12.5.5. Pharmacodynamic and Biomarker

#### **Pharmacodynamic**

#### PIP3 Peak Area Proportion for Sputum Sample

- PIP3 is the analyte of primary interest for the phospholipid data in sputum/Whole Blood, and Peak Area
  data from the mass spectrometer is the endpoint of interest. However, it is acknowledged that there will be
  some degree of variability between sputum/Whole blood samples due to differences in cell counts, and
  therefore it is favoured to first normalise PIP3 Peak Area values for each sample (by PIP2 Peak Area and
  PIP3 Peak Area); prior to analysis.
- More specifically the parameter of interest is: PIP3 Peak Area proportion.
   PIP3 Peak Area proportion is calculated from PIP2 Peak Area and PIP3 Peak Area, as follows:

$$PIP3$$
  $Peak$   $Area$   $proportion = \frac{PIP3 \ Peak \ Area}{PIP2 \ Peak \ Area} + PIP3 \ Peak \ Area$ 

- Evaluability was also assessed by the vendor based on sample outputs being above QC instrumentation criteria. Any non-evaluable data (as indicated in the database BIDEVCD=F) will be flagged and excluded from any summaries and analyses.
- PIP3 Peak Area, PIP2 Peak Area and, PIP3 Peak Area proportion, will be summarised by treatment group and study day

#### PIP3 For Peak Area Proportion for Whole Blood Sample

PBMCs isolated from whole blood and split 4 ways: -

- Unstimulated+DMSO (this is an unstimulated sample with the vehicle DMSO added)
- Unstimulated+NEMI (this is an unstimulated sample incubated with NEMI)
- Stimulated+DMSO (this is a sample stimulated with CD3+CD28 with the vehicle DMSO added)
- Stimulated+NEMI (this is a sample stimulated with CD3+CD28 and incubated with NEMI)

Individual Subject level Ratio for each of the below list group will be calculated for PIP3 Area proportion parameter for each of the timepoint separately

- Unstimulated+DMSO / Stimulated+DMSO
- Unstimulated+DMSO / Unstimulated+NEMI
- Stimulated+DMSO / Stimulated+NEMI

Note: PIP 3 Peak Area Proportion will be calculated separately for each of the above processing types.

#### Exploratory phospho-protein biomarkers(pAKT, AKT)

Individual Subject level Ratio for each of the below list group will be calculated for each parameter for each of the timepoint separately

- Unstimulated+DMSO / Stimulated+DMSO
- Unstimulated+DMSO / Unstimulated+NEMI
- Stimulated+DMSO / Stimulated+NEMI

204745

#### 12.5.6. **Efficacy**

#### **Efficacy**

#### Episodes of pulmonary and/or ear and sinus infections requiring anti- microbial treatment

Episodes of pulmonary and/or ear and sinus infections requiring anti- microbial treatment will be programmatically identified as follows:

- 1. Adverse Event dataset will be reviewed to identify any pulmonary and/or ear and sinus infections
  - If no AEs of pulmonary and/or ear and sinus infections were recorded, then no pulmonary and/or ear and sinus infections requiring anti- microbial treatment will be reported.
  - If AEs of pulmonary and/or ear and sinus infections were recorded, then proceed to step 2
- 2. A list of all concomitant medication (i.e. CONMEDS dataset with duplicated removed) will be sent to the Medical Monitor to identify and flag any anti-microbial treatments
  - If no anti-microbial treatments were identified, then no pulmonary and/or ear and sinus infections requiring anti- microbial treatment will be reported.
  - If anti-microbial treatments were identified, then proceed to step 3
- 3. Compare each pulmonary and/or ear and sinus infections AE with anti-microbial treatments concomitant medication
  - if antimicrobial treatment was taken within 7 days of the pulmonary and/or ear and sinus infections AE, then record as a pulmonary and/or ear and sinus infections requiring antimicrobial treatment

else no pulmonary and/or ear and sinus infections requiring anti- microbial treatment will be reported

204745

## 12.6. Appendix 6: Reporting Standards for Missing Data

# 12.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as subject who has completed all phases of the study including the follow-up visit.</li> <li>Withdrawn subjects were not replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

## 12.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| Soluble proinflammatory mediators | <ul> <li>Any values below the Lower Limit of Quantification (LLQ) will be assigned a value<br/>of ½ LLQ for display purposes in Figures and for computation of summary<br/>statistics.</li> </ul> |
| | <ul> <li>Any values above the Upper Limit of Quantification (ULQ) will be assigned to the ULQ for display purposes in Figures and for computation of summary statistics.</li> <li>Where biomarker concentrations are from an assay of an increased dilution factor the LLQ and ULQ will be multiplied by this factor.</li> <li>Note: Values sent to biostatistics team are already adjusted for this dilution factor Imputed values will be used in tables and figures, unless the proportion of imputed values at a given time point is large, in which case the summary statistics may not be presented for that time point and/or alternative actions will be taken and documented in the study report.</li> </ul> |
| | <ul> <li>Where values are imputed, the number of such imputations will be included as a<br/>summary statistic in the relevant summary tables.</li> </ul> |
| Plasma and BAL Urea Data | BLQ values will be imputed with the relevant (plasma or BAL fluid) LLQ divided by 2 • for the purpose of deriving the Dilution Factor. |
| Phospholipid<br>Data(PIP2,PIP3) | There is no quantifiable value for the LLQ for the phospholipid data. However, data with a particularly high noise/signal ratio will be deemed non evaluable by the external vendor. A flag for evaluability will be included in the listings and non-evaluable subjects will be excluded from summaries and analyses. |

204745

# 12.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail | |
|---|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. | |
| Adverse<br>Events | <ul> <li>Imputations in the adverse events dataset are used for slotting events to the appr<br/>study time periods and for sorting in data listings.</li> <li>Partial dates for AE recorded in the CRF will be imputed using the following convergence.</li> </ul> | |
| | Missing start day | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> </ul> </li> </ul> |
| | | <ul> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> |
| | Missing start day and month | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> </ul> |
| | Missing stop day | Last day of the month will be used. |
| | Missing stop day and month | No Imputation |
| | Completely missing start/end date | No imputation |
| | <ul> <li>Completely missin</li> </ul> | g start or end dates will remain missing, with no imputation applied. |
| Concomitant<br>Medications | Partial dates for ar<br>the following converge. | ny concomitant medications recorded in the CRF will be imputed using ention: |
| | Missing start day | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | Missing start day and month | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> </ul> |
| | Missing end day | A '28/29/30/31' will be used for the day (dependent on the month and year) |

204745

| Element | Reporting Detail | |
|---|---|---|
| | Missing end day and month | A '31' will be used for the day and 'Dec' will be used for the month. |
| | Completely missing start/end date | No imputation |
| | The recorded parti | al date will be displayed in listings. |

204745

# 12.7. Appendix 7: Values of Potential Clinical Importance

# 12.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Hematocrit | Ratio of | Male | 0.33 | 0.65 |
| Hematochi | 1 | Female | 0.33 | 0.65 |
| Haemoglobin | g/L | | 115 | 175 |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 600 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | 55 |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | | 40 | 120 |
| Glucose (Non-fasting) | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 155 |

| Liver Function | | | |
|--------------------|--------|----------|-------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2X ULN |
| AST/SGOT | U/L | High | ≥ 2X ULN |
| AlkPhos | U/L | High | ≥ 2X ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5X ULN |
| | µmol/L | | ≥ 1.5X ULN T. Bilirubin |
| T. Bilirubin + ALT | | High | |
| | U/L | | ≥ 2X ULN ALT |

204745

# 12.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTcF Interval | msec | | ≥ 500 |
| Absolute PR Interval | msec | < 100 | >240 |
| Absolute QRS Interval | msec | < 80 | > 120 |
| HR (Ventricular rate) | bpm | < 35 | >100 |
| Change from Baseline | Change from Baseline | | |
| Increase from Baseline QTc | msec | | ≥ 60 |

# 12.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------------|------------------------|--------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | <80 | >160 |
| Diastolic Blood Pressure | mmHg | ≤ 40 | ≥ 100 |
| Heart Rate | bpm | ≤ 40 | ≥ 100 |
| Temperature | °C | ≤35.5 | ≥ 37.5 |
| Respiration rate | breaths/min | ≤ 8 | ≥ 20 |

204745

#### 12.8. Appendix 8: Data Output Framework

To ensure transparent reporting of this study we have considered a decision framework in line with the study objectives outlined in Section 2.2.

- Original aim (primary endpoint) was to understand safety of PI3Kd inhibition in these
  patients. It was unknown at the time what would happen when turning the kinase off
  in an activated mutation state. Safety has been reviewed in stream, with no limiting
  effects observed.
- Secondary endpoint was PK. It is key to show similar (<2-fold) difference in PK vs COPD to be convinced of lung exposure.
- Exploratory endpoints are target engagement (PIP3), and downstream pharmacology (inflammatory cytokines)
- Team would want to see >30% reduction in PIP3 and >30% reduction in cytokines to be convinced of drug action in these patients.
- Team have significant experience in measuring PIP3 to show target engagement and have confidence in this readout.
- Team also have significant experience in lung cytokine measurement and feel this is higher risk due to variability. However, the inflammation should be entirely PI3Kddependent.

Thus the APDS Study Minimum Thresholds are as follows:

| Endpoint | APDS Study Minimu | um Thresholds | |
|---|---|---|---|
| Safety | Safety reviewed in stream, with no limiting AEs reported (n=4). No | | |
| (Primary) | cough to date, but po | st-inhalation wheeze i | reported in one subject |
| | Comparable Existing table | NEMI exposure(C <sub>tau</sub> ) | data is listed in below |
| | table | Existing NEMI<br>exposure<br>C <sub>tao</sub> (pg/mL) value | Interval for Geo. |
| PK | Day 1: 24h Post-<br>dose | 166 | (83, 332) |
| (Secondary) | Day 14: Pre-dose | 687 | (344,1374) |
| | Day 83: Pre-dose | 528 | (264,1056) |
| | Plasma Ctrough of | ed to indicate whether<br>concentration is at part<br>mparable <2 fold diffe | icular timepoint mentioned |
| Sputum PIP3 (Exploratory: Target Engagement) | >30% reduction PIP3 | B proportion from base | line |
| Sputum Cytokines<br>(Exploratory: Downstream<br>Pharmacology) | >30% reduction from | baseline IL-8, IL-6, TI | NFα, MMP9 |
| PIP3 in PBMCs | PIP3 in PBMCs | | |
| (Exploratory: Confirmation of patient | <ul> <li>&gt;30% inhibition (of unstimulated)</li> </ul> | | |
| sensitivity to PI3Kδ Inhibition) | <ul> <li>&gt;50% inhibition</li> </ul> | n (stimulated) | |

204745

# 12.9. Appendix 9: Abbreviations & Trade Marks

# 12.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| ELF | Epithelial lining fluid |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

204745

## 12.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| DISKUS |
| ELLIPTA |
| HARP |
| RANDALL NG |

Trademarks not owned by the GlaxoSmithKline Group of Companies [SAS]

204745

#### 12.10. Appendix 10: List of Data Displays

#### 12.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|-------------------------------|-------------|------------|
| Study Population | 1.1 to 1.10 | |
| Efficacy | 2.1 to 2.2 | |
| Safety | 3.1 to 3.12 | |
| Pharmacokinetic | 4.1 to 4.4 | |
| Pharmacodynamic and Biomarker | 6.1 to 6.11 | 6.1 to 6.6 |
| Section | Listi | ngs |
| ICH Listings | 1 to | 29 |
| Other Listings | 30 to | 41 |

## 12.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock shells for Data Displays

| Section | Figure | Table | Listing |
|-------------------------------|--------|--------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic and Biomarker | PD_Fn | PD_Tn | PD_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 12.10.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

204745

# 12.10.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1.1. | All Subjects | ES1 | Summary of Participant Disposition for the Participant Conclusion Record | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | All Subjects | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC |
| Protoc | ol Deviation | | | | |
| 1.4. | All Subjects | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| Demog | raphic and Bas | seline Characteris | tics | | |
| 1.5. | All Subjects | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC |
| 1.6. | All Subjects | DM11 | Summary of Age Ranges | EudraCT | SAC |
| 1.7. | All Subjects | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |
| Popula | tion Analysed | | | | |
| 1.8. | Screened | SP1 | Summary of Study Populations | Summarize by each treatment group (i.e. NEMI 1000mcg Diskus, NEMI 700mcg Ellipta, NEMI 500mcg Ellipta) and ALL NEMI, No Treatment group Refer to Table 1.6 in gsk2269557/mid201928/final_01 | SAC |
| Prior a | Prior and Concomitant Medications | | | | |
| 1.9. | All Subjects | CM1 | Summary of Concomitant Medications | ICH E3 | SAC |

204745

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Exposui | Exposure and Treatment Compliance | | | | |
| 1.10. | All Subjects | EX1 | Summary of Exposure to Study Treatment | | SAC |

# 12.10.5. Efficacy Tables

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| FEV1 | | | | | |
| 2.1. | All Subjects | PFT1 | Summary of Absolute FEV1 (L) Data | Refer PII115119/ Part_A /Table 3.18<br>Add footnote "Note: Maximum value of<br>the three readings has been used." | SAC |
| 2.2. | All Subjects | PFT3 | Summary of Change from Baseline FEV1 (L) Data | Refer PII115119/ Part_A /Table 3.19 | SAC |

204745

# 12.10.6. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events (AEs) | | | | • |
| 3.1. | All Subjects | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.2. | All Subjects | AE1 | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.3. | All Subjects | AE15 | Summary of Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Required by Register Disclosure for FDAAA and EudraCT. | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | 1 |
| 3.4. | All Subjects | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | SAC |
| 3.5. | All Subjects | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | IDSL | SAC |
| Labora | tory: Chemistr | y | | | |
| 3.6. | All Subjects | LB1 | Summary of Chemistry Changes from Baseline | ICH E3 | SAC |
| Labora | Laboratory: Hematology | | | | |
| 3.7. | All Subjects | LB1 | Summary of Hematology Changes from Baseline | ICH E3 | SAC |
| Labora | tory: Hepatobil | liary (Liver) | | | |
| 3.8. | All Subjects | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | SAC |

204745

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.9. | All Subjects | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | SAC |
| ECG | | | | | |
| 3.10. | All Subjects | EG1 | Summary of ECG Findings | IDSL | SAC |
| 3.11. | All Subjects | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC |
| Vital Si | Vital Signs | | | | |
| 3.12. | All Subjects | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | SAC |

# 12.10.7. Pharmacokinetics Table

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Plasma | PK | | | | |
| 4.1. | PK | PK01 | Summary of Plasma Nemiralisib Pharmacokinetic Concentration-Time Data | | SAC |
| 4.2. | PK | PK_T1 | Summary of Log-Transformed Plasma Nemiralisib Pharmacokinetic Concentration - Time Data (pg/mL) | Include flag derived for minimum threshold criteria as mentioned in Section 12.8. | SAC |
| Lung e | Lung epithelial lining fluid (ELF) and Bronchoalveolar lavage (BAL) | | | | |
| 4.3. | PK | PK_T2 | Summary of Urea Dilution Factor Data | | SAC |
| 4.4. | PK | PK_T3 | Summary of Derived Lung ELF and Cell Pellet Nemiralisib Pharmacokinetic Concentrations and Volume Data | | SAC |

204745

# 12.10.8. Pharmacodynamic and Biomarker Tables

| Phar | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| PIP2 | PIP2/PIP3 | | | | |
| 6.1. | All Subjects | PD_T1 | Summary of Phospholipid Data (Absolute) in Sputum | | SAC |
| 6.2. | All Subjects | PD_T3 | Summary of Phospholipid Data (Change from Baseline) in Sputum | Includes only PIP3 Proportion parameter | SAC |
| 6.3. | All Subjects | PD_T2 | Summary of Phospholipid Data (Absolute) in Blood | | SAC |
| 6.4. | All Subjects | PD_T4 | Summary of Phospholipid Data (Change from Baseline) in Blood | Includes only PIP3 Proportion parameter | SAC |
| 6.5. | All Subjects | PD_T5 | Summary of statistical analysis of Loge transformed PIP3 Area Proportion | Refer Table 2.62 in 201928/final_02 RE | SAC |
| Solul | ble Proinflamm | atory Mediators | | | |
| 6.6. | All Subjects | PD_T6 | Summary Statistics (Absolute): Soluble proinflammatory mediators | Includes IL-8, IL-6, TNFa & MMP9 | SAC |
| 6.7. | All Subjects | PD_T6 | Summary Statistics (Change from Baseline): Soluble proinflammatory mediators | Includes IL-8, IL-6, TNFa & MMP9 | SAC |
| 6.8. | All Subjects | PD_T7 | Summary Statistics (Log-Transformed Absolute): Soluble proinflammatory mediators | Includes IL-8, IL-6, TNFa & MMP9 | SAC |
| 6.9. | All Subjects | PD_T7 | Summary Statistics (Log-Transformed Change from Baseline): Soluble proinflammatory mediators | Includes IL-8, IL-6, TNFa & MMP9 | SAC |
| Immu | une cell and Ly | mphocyte cell subs | sets | | |
| 6.10. | All Subjects | LB1 | Summary of Blood Lymphocyte Cell Subsets (Change from Baseline) | Include Blood Sample type data only | SAC |
| Phos | Phospho-protein biomarkers(pAKT,AKT) | | | | |
| 6.11. | All Subjects | PD_T2 | Summary of Phospho-protein Biomarkers (Absolute) | Include Sample type (i.e. Sputum, BAL etc) as Page by Variable Include pAKT ,AKT parameter | SAC |

204745

# 12.10.9. Pharmacodynamic and Biomarker Figures

| Pharm | Pharmacodynamic and Biomarker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| PIP2, F | PIP3 | | | | |
| 6.1. | All Subjects | PD_F1 | Individual subjects profile plot of Phospholipid Data in Sputum | Different colour legend for each subject . Ignore processing type panel in mock shell for Sputum data. Page by Parameter (PIP2,PIP3,PIP3 proportion) | SAC |
| 6.2. | All Subjects | PD_F2 | Geometric Mean and 95% Confidence Interval for Phospholipid Data in Sputum | Different colour legend for each parameter | SAC |
| 6.3. | All Subjects | PD_F1 | Individual subjects profile plot of Phospholipid Data in Blood | Page by Parameter (PIP2, PIP3, PIP3 proportion) Different colour legend for each subject Different plot of processing type and (1st page include 4 different processing type and 2nd page is for 3different processing type comparison values) | SAC |
| 6.4. | All Subjects | PD_F2 | Geometric Mean and 95% Confidence Interval for Phospholipid Data in Blood by Processing Type | Different colour legend for each processing type 1st page include figure having 4 different line for each processing type estimates and 2nd plot is for 3different processing type comparison values) | SAC |
| Phosp | ho-protein bion | narkers(pAKT,AK | T) | | |
| 6.5. | All Subjects | PD_F1 | Individual subjects profile plot for phospho-protein biomarkers Data in Blood | Different plot of processing type and (1st page include 4 different processing type and 2nd page is for 3 different processing type comparison values) | SAC |
| 6.6. | All Subjects | PD_F2 | Geometric Mean and 95% Confidence Interval for phospho-protein Biomarkers in Blood by Processing Type | Different colour legend for each processing type 1st page include figure having 4 different line for each processing type estimates and 2nd plot is for 3different processing type comparison values) | SAC |

204745

# 12.10.10. ICH Listings

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | Subject Disposition | | | | |
| 1. | Screened | ES6 | Listing of Reasons for Screen Failure | | SAC |
| 2. | Screened | ES9 | Listing of Subjects Who Were Rescreened | | SAC |
| 3. | All Subjects | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 4. | All Subjects | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC |
| 5. | All Subjects | TA1 | Listing of Planned and Actual Treatments | IDSL | SAC |
| Protoc | ol Deviations | 1 | | | <b>-</b> |
| 6. | Screened | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 7. | All Subjects | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Popula | tions Analysed | 1 | | | <u>.</u> |
| 8. | Screened | SP3 | Listing of Participants Excluded from Any Population | | SAC |
| Demog | raphic and Ba | seline Characteris | etics | | |
| 9. | All Subjects | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 10. | All Subjects | DM9 | Listing of Race | ICH E3 | SAC |
| Prior a | Prior and Concomitant Medications | | | | |
| 11. | All Subjects | CM3 | Listing of Concomitant Medications | IDSL | SAC |
| 12. | All Subjects | POP_L1 | Listing of Ear, Sinus and Pulmonary Infection History over Previous Two Years | | SAC |

204745

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Expos | ure and Treatm | ent Compliance | | | |
| 13. | All Subjects | EX3 | Listing of Exposure Data | ICH E3 | SAC |
| Advers | se Events | | | | |
| 14. | All Subjects | AE8 | Listing of All Adverse Events | ICH E3 | SAC |
| 15. | All Subjects | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| 16. | All Subjects | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Seriou | s and Other Sig | nificant Adverse | Events | | |
| 17. | All Subjects | AE8 | Listing of Serious Adverse Events | ICH E3 Include a column to flag fatal and non-fatal SAEs | SAC |
| 18. | All Subjects | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |
| 19. | All Subjects | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| Hepato | biliary (Liver) | | | | |
| 20. | All Subjects | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | SAC |
| 21. | All Subjects | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | SAC |
| 22. | All Subjects | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | SAC |
| All Lab | oratory | | | | |
| 23. | All Subjects | LB5 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| 24. | All Subjects | LB5 | Listing of Laboratory Values of Potential Clinical Importance | | SAC |
| 25. | All Subjects | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |

204745

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 26. | All Subjects | UR2 | Listing of Urinalysis Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| ECG | | | | | |
| 27. | All Subjects | EG3 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| 28. | All Subjects | EG5 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | SAC |
| Vital Signs | | | | | |
| 29. | All Subjects | VS4 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |

204745

# 12.10.11. Non-ICH Listings

| Non-IC | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Pharm | nacokinetic | | | | |
| 30. | PK | PK07 | Listing of Plasma Nemiralisib Concentration-time Data | | SAC |
| 31. | PK | PK_L1 | Listing of Plasma Urea and BAL Fluid Urea Data | | SAC |
| 32. | PK | PK_L2 | Listing of BAL Fluid and Derived Lung ELF Nemiralisib Pharmacokinetic Concentration Data | | SAC |
| Pharm | acodynamic (P | IP2/PIP3) | | | |
| 33. | All Subjects | PD_L1 | Listing of Phospholipid Data in Sputum | | SAC |
| 34. | All Subjects | PD_L2 | Listing of Phospholipid Data in Blood | | SAC |
| Pharm | acodynamic (S | oluble proinflamn | natory mediators) | | |
| 35. | All Subjects | PD_L3 | Listing of Individual Subject Soluble proinflammatory mediators Data | Refer PII115119/Part A/Listing 34 | SAC |
| Pharm | acodynamic (In | nmune cell and L | ymphocyte cell subsets) | | |
| 36. | All Subjects | PD_L4 | Listing of Immune Cell Count Data | | SAC |
| 37. | All Subjects | PD_L4 | Listing of Lymphocyte cell subsets | | SAC |
| Pharm | acodynamic (p | AKT/AKT) | | | |
| 38. | All Subjects | PD_L6 | Listing of Phospho-protein biomarkers | | SAC |
| Pharm | acodynamic (A | ntibody Level) | | | |
| 39. | All Subjects | PD_L5 | Listing of Antibody Level | | SAC |
| Efficac | y . | | | | • |
| 40. | All Subjects | PFT8 | Listing of FEV1 (L) Data | | SAC |
| 41. | All Subjects | EFF_L1 | Listing of Episodes of Pulmonary and/or Ear and Sinus Infections Requiring Anti-Microbial Treatment | | SAC |

204745

# 12.11. Appendix 11: Example Mock shells for Data Displays

Data Display Specification will be made available on request